CLINICAL TRIAL: NCT04441463
Title: Simultaneous Study of the Serum Tryptase Level of the Mother and the Child During Childbirth
Brief Title: Simultaneous Study of the Serum Tryptase Level of the Mother and the Child During Childbirth (TryPla)
Acronym: TryPla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2020 PONS; 2020-A01526-33 (Other: ANSM)
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Newborn; Parturient
Keywords: Tryptase; Neonatal; Newborn; Transplacental passage; Mast cell; Inflammation; Biomarker
MeSH Terms: conditions — Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohort (Experimental): Mother-child couple
  Interventions: Biological: Blood sampling for tryptase analysis

INTERVENTIONS:
Biological: Blood sampling for tryptase analysis — 3 bloods test
  * One blood sample taking from the mother's vein punction, during the delivery.
  * One blood sample tanking from umbilical cord.
  * One blood sample taking from the baby in day 3 of life, during the Guthrie test.

SUMMARY:
Currently the neonatal serum level of severals proteins can be used as an indicator of subsequent risk. For example, we plan to explore the neonatal kinetics of tryptase and other immune proteins as potential markers for the risk of postnatal complications, particularly in premature babies. However, today no study has shown whether the tryptase level in the newborn is a reflection of fetal synthesis alone, or that of the mother by possible transplacental passage. There is also no database that has defined normal values for tryptase in cord blood.

Our main objective is to determine the correlation between the level of maternal tryptase and that of the newborn in cord blood immediately after birth in order to estimate the transplacental passage of this molecule.

DETAILED DESCRIPTION:
* The protocole will be explain to the family in delivery room, an information note will be given, and we will let the time to think about it.
* In a second time investigator will make the mother sign a consent, that participant could retract any time then.
* A blood sample will be taken from the mother within 2 hours of delivery, using a standard blood test.
* A sample will be taken from the infant by blood drawn from the umbilical cord (non-invasive and painless sample).
* A final blood sample from your newborn will be collected at the time of the Guthrie test (systematic screening for congenital diseases) already scheduled for the new born on the third day of life.
* This blood sample will be sent to the immunology laboratory of the Clermont-Ferrand University Hospital where specific biological assays will be carried out.
* Blood samples will be stored for future use in studies.
* A collection of data concerning the child, childbirth and the results of biological analyzes will be carried out. All data will be coded.
* A phone call will be made at 3 months of life, to review the state of the child's health during his first months of life.

ELIGIBILITY:
Inclusion Criteria:

* Mother-child couple
* Childbirth at the Clermont-Ferrand University Hospital.
* Affiliated to a social security system

Exclusion Criteria:

* Newborns whose holders of parental authority are protected by law (under guardianship, placed under the protection of justice)
* Newborns whose holders of parental authority are under the age of 18
* Fetal pathology, excluding prematurity.
* emergency caesarean section, because o life threatening condition for the fetus or the mother.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Rate of blood tryptase | at birth (day 0)
  blood sample for biomarker reflecting the mast cell activity

SECONDARY OUTCOMES:
Rate of blood tryptase | day 3
  blood sampling for biomarker reflecting the mast cell activity
Incidence of infectious disease and hospitalization | Month 3
  call phone for evaluation of medical condition for child by questionnaire about physical history in the past 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Maguelonne Pons, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France